CLINICAL TRIAL: NCT00210756
Title: Comparative Pharmacokinetic and Pharmacodynamic Study of Epoetin Alfa (PROCRIT) in Anemic Critically Ill Patients Randomized to One of Six Dose Regimens for 15 Days
Brief Title: Pharmacokinetic/ Pharmacodynamic Study of Epoetin Alfa (PROCRIT) in Critically Ill Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004603
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Critical Illness
Keywords: Anemia; pharmacokinetics; erythropoetin; Epoetin alfa; erythropoetin recombinant; Critical care; critical illness, intensive care,
MeSH Terms: conditions — Anemia; Critical Illness | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to describe the pharmacokinetics (PK) of six different dosing regimens of epoetin alfa (PROCRITÂ®) in anemic critically ill subjects

DETAILED DESCRIPTION:
Currently, the optimal dosing regimen for achieving and maintaining target Hb concentrations in various clinical settings remains incompletely defined. Both IV and SC routes of administration are used in the clinical setting and have been shown to be effective despite different bioavailability and pharmacokinetic profiles. This study is designed to describe the pharmacokinetic and pharmacodynamic profiles of several different epoetin alfa dosing regimens administered by both IV and SC routes in anemic critically ill patients admitted to a critical care area. The dosing regimens selected will be compared among themselves and against the 40,000 IU SC weekly dosing regimen (A) being used in a large registration trial. Specifically, the six dosing regimens were selected to gather PK and PD data about the following questions: 1) Will an early large Cmax, achieved by IV dosing, stimulate more reticulocytosis? (IV vs. SC dosing regimens A vs. B, C vs. D, E vs. F); 2) Do smaller more frequent doses of the same total dose result in the same PD profile? (A vs. C, B vs. D); 3) Does an IV load improve PD response? (E and F vs. C and D); 4) Do large frequent loading doses accumulate? (A vs. E and B vs. F). Results of this study will provide a pharmacokinetic foundation for understanding and potentially maximizing the pharmacodynamic effects of different dosing options in the critically ill patient. In order to maximize subject safety, all dosing will cease when subject's hemoglobin is > 13g/dL. Group A:40 K SC Qw: Days 1,8,15; Group B:40 K IV Qw: Days 1,8,15; Group C:15 K SC QOD: Days 1,3,5,7,9,11,13,15; Group D:15 K IV QOD: Days 1,3,5,7,9,11,13,15; Group E:40 K SC Days 1 and 3, then 15 K SC QOD: Days 5,7,9,11,13,15; Group F: 40 K IV Days 1 and 3, then 15 K SC QOD: Days 5,7,9,11,13,15

ELIGIBILITY:
Inclusion Criteria:

* Critically ill subject admitted to a critical care area with a medical diagnosis, (non-surgical, non-trauma) and without evidence of acute blood loss
* or Critically ill subject who develops a medical diagnosis after surgery or trauma and who has no evidence of active bleeding within the prior week and no current transfusion needs
* Expected hospital stay of >= 7 days beyond study entry, age >=18 years
* Hb:<=12 g/dL.

Exclusion Criteria:

* Primary admitting diagnosis to the critical care area of acute ischemic cardiac disease or ischemic neurological disease (including but not limited to myocardial infarction or unstable angina, transient ischemic attack, cerebrovascular event)
* History of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* Iron deficiency (defined as serum ferritin <50 micrograms/L)
* History of untreated chronic B12 or Folate deficiency (e.g. pernicious anemia). Patients with B12 and folate deficiencies being treated currently may enter the study
* Renal failure on dialysis, including continuous renal replacement therapy (CRRT), at the time of enrollment
* Evidence of acute blood loss within 1 week of enrollment or an active diagnosis of acute or chronic blood loss or hemolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-02; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to describe the PK profiles of six different dosing regimens of epoetin alfa in anemic critically ill subjects, including regimen A, that is being used in a large registration trial

SECONDARY OUTCOMES:
To determine reticulocyte response (absolute and %) to the six dosing regimens, as well as the Hb, Hct, and RBC count response. Compare the PD profiles of each dosing regimen to dosing regimen A. describe the safety profile of the six dosing regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Comparative Pharmacokinetic and Pharmacodynamic Study of Epoetin Alfa (PROCRIT) in Anemic Critically Ill Patients Randomized to One of Six Dose Regimens for 15 Days. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=605&filename=CR004603_CSR.pdf